CLINICAL TRIAL: NCT06297551
Title: Prospective Study of Leukemia Stem Cells Fractional Change in Peripheral Blood and Its Correlation With Therapeutic Outcome in Acute Myeloid Leukemia
Brief Title: Acute Myeloid Leukemia and Markers of Leukemia Stem Cells (CLL1 and CD45RA)
Status: Recruiting | Type: Observational
Sponsor: Suhu Liu (Other)
Responsible Party: Sponsor-Investigator, Suhu Liu, Assistant Professor of Medicine, Stony Brook University
Organization: Stony Brook University (Other)
Other Study IDs: SBU-AML-LSC; IRB2023-00528 (Other: Stony Brook University)
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Quantification of blood cells positive for CLL1 and CD45RA surface markers by flow cytometry — During induction therapy for AML, researchers will measure the relative percentage of hematopoietic stem cells (defined by markers CD34+/CD38-) that test positive for CLL1 and CD45RA surface markers in the blood of participants on day 3, 5 and 7 days of systemic therapy. The variation of blood cells positivity for these markers, will be correlated with treatment outcome (complete response, partial response, no response), as determined by a bone marrow biopsy done approximately 4 weeks after induction chemotherapy.

SUMMARY:
Acute myeloid leukemia (AML) is a malignant disorder of the bone marrow and the most common form of acute leukemia in adults. Patient with AML have the shortest survival compared to other forms of leukemia. In the past 6 years, several new therapies have been approved.

Biomarkers are in urgent need to guide therapeutic regimen selection in order to maximize the benefit of available therapies and minimize treatment toxicity. Current standard practice is to perform bone marrow biopsy at end of treatment cycle (each cycle around 28 days), and based on bone marrow finding, to decide further treatment plan. It is invasive and time consuming.

In this study investigators will study whether tracking leukemia stem cells (LSC) in peripheral blood during early treatment cycle may provide a non-invasive method to predict therapeutic outcome at end of treatment cycle. A retrospective study found that LSC fractional change, defined by two LSC markers, named CLL1 and CD45RA, is highly correlated with therapeutic outcome. Further more, CLL1 and CD45RA positive LSC fraction demonstrates a high concordance between bone marrow and peripheral blood, offering the opportunity to track CLL1 and CD45RA positive LSC fraction non-invasively in peripheral blood during treatment.

This pilot study will allow the investigators to decide whether testing CLL1 and CD45RA positive LSC in peripheral blood during leukemia treatment is feasible in clinical practice. This result will lay the foundation for designing future trials using CLL1 and CD45RA positive LSC fractional change to optimize therapeutic strategy for patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute myeloid leukemia
* ability to receive treatment for acute myeloid leukemia at the research center
* elevated values of CLL1A and CD45RA positive cells at the time of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with acute myeloid leukemia, undergoing systemic chemotherapy (high or low intensity)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between the relative fraction of Leukemia Stem Cells (LSC) vs Hematopoietic Stem Cells (HSC) and treatment response | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suhu Liu, MD PhD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No